CLINICAL TRIAL: NCT00881842
Title: Immunogenicity, Reactogenicity and Safety of the Trivalent Influenza Subunit Vaccine Influvac® for the Season 2009/2010. An Open-Label, Baseline-Controlled Multi-Center Study in Two Groups: Adult Subjects and Elderly Subjects
Brief Title: Annual Study to Investigate Inactivated Subunit Influenza Vaccine Due to New Virus Strains for the 09/10 Season
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Biologicals (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Organization: Abbott (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: S201.3.128; 2009-010900-27 (EudraCT Number)
Record Dates: First submitted 2009-04-14; First posted 2009-04-15 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Influenza
Keywords: Influenza; Vaccine; CHMP criteria
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: Trivalent influenza subunit vaccine Influvac

INTERVENTIONS:
Biological: Trivalent influenza subunit vaccine Influvac — 3x 15mcg HA per 0.5 ml,trivalent one injection at Day 1

SUMMARY:
Influenza (flu) viruses change continuously, therefore also the parts of viruses used in influenza vaccines can vary from year to year. In Europe, manufacturers/marketing holders of these vaccines are required to be involved in ongoing clinical trials and to present the results to the competent authorities each year. The current study is a phase IIIa clinical trial with a commercially available vaccine (Influvac®) supplied in pre filled syringes. It is part of the ongoing clinical trial program for Influvac® and will be done to assess the immunogenicity and safety and tolerability of next season's trivalent influenza subunit vaccine in two groups of subjects in good health: subjects aged >= 18 and <= 60 years and subjects >= 61 years of age (elderly).

ELIGIBILITY:
Inclusion Criteria

* Willing and able to give informed consent and able to adhere to all protocol required study procedures.
* Men and women aged >= 18 and <= 60 years or >= 61 years of age at the day of study vaccination.
* Being in good health as judged by medical history, physical examination and clinical judgment of the investigator.

Exclusion Criteria

* Known to be allergic to eggs, chicken protein, gentamicin or any other constituent of the vaccine.
* A serious adverse reaction after a previous (influenza) vaccination.
* Presence of any significant condition that may prohibit inclusion as determined by the investigator.
* Having received vaccination against influenza within the previous six months before study vaccination or planned vaccination during the study period.
* A history of Guillain-Barré syndrome or active neurological disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
HI titers and its derived parameters after 2 weeks (seroprotection, seroconversion and mean fold increase), reactogenicity and inconvenience of Influvac® 2008/2009 as defined by the CHMP guideline for influenza vaccines. | 2 weeks
HI titers and its derived parameters after 3 weeks (seroprotection, seroconversion and mean fold increase), reactogenicity and inconvenience of Influvac® 2008/2009 as defined by the CHMP guideline for influenza vaccines. | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hanka de Voogd, MD, Study Director — Abbott Healthcare Products B.V
Locations (2):
- Site Reference ID/Investigator# 59243, Tessenderlo, Belgium
- Site Reference ID/Investigator# 59244, Hamburg, Germany